CLINICAL TRIAL: NCT03353896
Title: Pilot Trial of NovoTTF -200A (TTFields) in Patients With Newly Diagnosed High Risk Oligodendrogliomas
Brief Title: NovoTTF-200A Device in Treating Patients With Newly Diagnosed High Risk Oligodendroglioma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6B-15-1; NCI-2017-02074 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EF-OLIGO-15; 6B-15-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Anaplastic Oligodendroglioma; Oligoastrocytoma; Oligodendroglioma
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (medical device) (Experimental): Beginning 4-8 weeks after standard of care treatment, patients wear NovoTTF-200A device over 18 hours QD. Treatment continues for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: Wear novoTTF-200A; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Device: Wear novoTTF-200A — Wear novoTTF-200A device
  Other Names: Medical Devices
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot clinical trial studies the side effects of NovoTTF-200A device in treating patients with newly diagnosed high risk oligodendroglioma. NovoTTF-200A device is a portable battery operated device which produces tumor treating (TT)Fields in the body by means of surface electrodes placed on the skin. TTFields are very low intensity, intermediate frequency electric fields that may slow the growth of tumor cells in patients with high risk oligodendroglioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the safety and tolerability of the TTFields treatment in patients with newly diagnosed high risk oligodendroglioma following standard of care treatment.

SECONDARY OBJECTIVES:

I. To estimate the proportion of patients who tolerated 75% of treatment goal at months 6, 12, 24.

II. To estimate the progression free survival time. III. To assess quality of life. IV. To assess whether or not there is a correlation between genomics and the efficacy of the TTFields treatment.

OUTLINE:

Beginning 4-8 weeks after standard of care treatment, patients wear NovoTTF-200A device over 18 hours daily (QD). Treatment continues for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 months and then monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed oligodendroglioma (oligo) (low grade oligo, low grade mixed oligoastrocytoma, anaplastic oligo, anaplastic mixed oligo) by histology and or molecular classification
* Surgically sub-total or unresectable tumors, i.e. in insula, including but not limited to the insula and received standard of care (SOC) radiation
* Historical pathological tissue evidence of high risk oligo (low grade oligo, low grade mixed oligoastrocytoma, anaplastic oligo, anaplastic mixed oligo) by histology and or molecular classification
* 1p and 19q deletion status known
* IDH 1 & 2 mutations status known
* MGMT status known
* Karnofsky equal or greater than 70
* Life expectancy at least 3 months
* Participants of childbearing age must use effective contraception

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Actively participating in another clinical treatment trial
* Tumor progression after radiation
* Pregnant
* Has implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain
* Documented clinically significant cardiac arrhythmias
* Infra-tentorial tumor

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of the NovoTTFields treatment in patients with high risk oligodendroglioma | Up to 2 months after treatment
  Number of patients with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chen, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States